CLINICAL TRIAL: NCT04899570
Title: A Prospective Phase II Study of Zanubrutinib Combined With R-CHOP in Newly-diagnosed Intravascular Large B-cell Lymphoma
Brief Title: Zanubrutinib Combined With R-CHOP in Newly-diagnosed Intravascular Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-008
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Intravascular Large B-Cell Lymphoma
Keywords: Intravascular Large B-Cell Lymphoma; zanubrutinib; R-CHOP
MeSH Terms: interventions — zanubrutinib; Rituximab; Cyclophosphamide; Epirubicin; Vindesine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib combined with R-CHOP (Experimental): The experimental arm will be treated zanubrutinib combined with R-CHOP regimen for 8 cycles. The interim evaluation will be performed after 4 cycles, and the patients who can't achieve PR or CR will be withdrawn from this trial and receive salvage regimens.
  After 8 cycles of ZR-CHOP, the patients will be followed for 2 years to evaluate the PFS.
  Interventions: Drug: Zanubrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vindesine; Drug: Prednisone

INTERVENTIONS:
Drug: Zanubrutinib — 160mg Bid, oral, d1-21 in a 21-day cycle for 8 cycles.
  Other Names: BRUKINSA
Drug: Rituximab — Rituximab 375mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 8 cycles will be prescribed as protocol
  Other Names: Rituxan
Drug: Cyclophosphamide — Cyclophosphamide 750mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 8 cycles will be prescribed as protocol
Drug: Epirubicin — Epirubicin 70mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 8 cycles will be prescribed as protocol
Drug: Vindesine — Vindesine 4mg intravenous infusion d1, every 21 days for 1 cycle. 8 cycles will be rescribed as protocol
Drug: Prednisone — Prednisone 60mg/m2 orally d1-5, every 21 days for 1 cycle. 8 cycles will be rescribed as protocol

SUMMARY:
This is a prospective single-arm phase II study, and the purpose of this study is to evaluate the efficiency of zanubrutinib combined with R-CHOP regimen in newly diagnosed primary intraocular lymphoma. Progression-free survival (PFS) of the cohort is the primary endpoint.

DETAILED DESCRIPTION:
All the eligible patients will be treated with ZR-CHOP regimen (Rituximab 375mg/m2 IV d1, cyclophosphamide 750mg/m2 IV d1, epirubicin 70mg/m2 IV d1, vindesine 4mg IV d1，prednison 60mg/m2 d1-5 PO). An interim evaluation will be performed after 4 cycles, the patients who achieve CR or PR will receive another 4 cycles of ZR-CHOP.

The patients with stable disease (SD) or progressed disease (PD) will withdraw from the trial and receive salvage regimens.

During the following-up, surveillance physical examination and CT scans should be performed every 6 months for 2 years to determine the status of disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteered to participate in the study and signed the Informed Consent
* Age ≥18 years old ≤70 Years old, male or female
* Expected survival ≥ 12 weeks
* Intravascular large B-cell lymphoma confirmed by cytology or histology according to WHO2016 criteria
* Never received any anti-tumor therapies.
* Adequate organ function and adequate bone marrow reserve

Exclusion Criteria:

* Malignant tumors other than IVLBCL within 5 years prior to screening, except cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery
* Active HIV, HBV, HCV or treponema pallidum infection
* Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need therapy
* Female subjects who have been pregnant or breastfeeding, or who plan to conceive during or within 1 year after treatment, or male subjects' partner plans to conceive within 1 year after their cell transfusion
* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | from the date of treatment to the subject finished his 2 years follow-up phase or the disease relapsed or the death due to lymphoma
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow up without relapsing.

SECONDARY OUTCOMES:
overall response rate(ORR) | 6 weeks after the end of 8 cycles of induction (each cycle is 21 days).
  ORR was calculated by the proportion of patients who achieved complete remission and partial remission.

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, Study Chair — Department of Hematology, Peking University First Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China